CLINICAL TRIAL: NCT01199614
Title: HEXT: The Hypoparathyroidism Studies, EXTended: The Effect of PTH on the Skeleton in Hypoparathyroidism
Brief Title: HEXT (Hypo EXTended): Effect of PTH on Skeleton in Hypoparathyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: NPS Pharma (Industry); Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAE0544
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; Hypopara; HPTH; Hypocalcemia; Hypercalciuria; PTH; PTH(1-84)
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia; Hypercalciuria | interventions — Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label PTH(1-84) (Experimental): open-label PTH(1-84) / variable dosing: 25mcg every other day, 25mcg every day, 50mcg every day, 75mcg every day, 100mcg every day
  Interventions: Drug: open-label PTH(1-84)

INTERVENTIONS:
Drug: open-label PTH(1-84) — open label PTH(1-84) at either 25mcg every other day, 25mcg every day, 50mcg daily, 75mcg daily, or 100mcg daily
  Other Names: rhPTH1-84; rhPTH(1-84); PTH1-84; PTH(1-84); PTH; parathyroid hormone

SUMMARY:
This is an open-label study of PTH(1-84) treatment that seeks:

1. To determine the actions of PTH(1-84) to provide long term control of serum calcium and urinary calcium excretion with use of standard amounts of calcium and vitamin D supplementation.
2. To determine the extent to which PTH(1-84) improves quality-of-life on long-term basis.
3. To establish the safety of PTH(1-84) when administered for up to 12 years.
4. To attempt to quantify improvements in the typical signs/symptoms of hypoparathyroidism post PTH administration.

There will be one visit conducted every six months in the study offices of the principal investigator, Dr. John Bilezikian. In addition to these visits, there will be, for new patients who have not used PTH (1-84) before, a Screening Visit four weeks prior to the baseline visit for the purpose of performing screening labs as well as a Pre-Baseline Local Quest Lab performed to ensure stability prior to Baseline.

DETAILED DESCRIPTION:
Hypoparathyroidism is a rare disorder in which parathyroid hormone (PTH) is markedly decreased or absent from the circulation. It is the only remaining hormone deficiency state for which replacement with the missing hormone has been heretofore unavailable. The hypoparathyroid state is due either to autoimmune destruction of the parathyroid glands or to loss of parathyroid function after neck surgery. Without PTH, calcium homeostasis is markedly abnormal, the most salient clinical feature of which is a reduced serum calcium concentration. The hypocalcemia is associated with other important abnormalities such as markedly reduced parameters of bone turnover. PTH(1-84) is the ideal therapeutic approach to hypoparathyroidism. The current mainstay of therapy, calcium and vitamin D, has important clinical limitations. Large doses of calcium and vitamin D are required and often associated with hypercalciuria and vitamin D toxicity. Moreover, this approach does not correct the skeletal deficiencies resident in the bones themselves due to lack of PTH. In contrast, PTH(1-84) replaces precisely what is missing in this disorder. The research question is: What are the long-term safety and efficacy parameters of PTH(1-84) therapy in hypoparathyroidism?

Preliminary data suggest that treatment with PTH(1-84) for up to 4 years improves control of the serum and urine calcium concentration safely. Since hypoparathyroidism is a chronic disorder, it is important to know whether these salutary effects continue to be seen beyond 4 years. There is a need to determine the safety and efficacy treatment of PTH(1-84) in hypoparathyroidism beyond 4 years.

ELIGIBILITY:
For Returning Participants or participants graduating from one of the parent studies:

Inclusion Criteria:

* Must have participated in and concluded the CL1-11-040, PAR-C10-007 or PAR-C10-008 Study at any site in the continental United States
* Must have participated in and concluded the Hypopara Study at Columbia University

Exclusion Criteria:

* failure to have completed either of the inclusionary studies

For New Participants (20 anticipated):

INCLUSION CRITERIA:

1. Signed and dated informed consent form (ICF) before any study-related procedures are performed.
2. Adult males or females 18 to 85 years of age.
3. History of hypoparathyroidism for ≥ 18 months, including evidence of hypocalcemia and concomitant serum intact PTH concentrations below the lower limit of normal within 12 months prior to Baseline.
4. Requirement for calcitriol ≥0.25 mcg per day per day prior to Baseline.
5. Requirement for supplemental oral calcium ≥ 1500 mg per day between supplemental and dietary sources.
6. Serum thyroid function tests within normal laboratory limits at screening for all subjects not receiving thyroid hormone replacement therapy. For patients on thyroid hormone replacement therapy, the dose must have been stable for at least 3 months prior to screening
7. serum creatinine < 1.5 mg/dL on a single measurement prior to use of study drug
8. Physically capable of performing daily subcutaneous (SQ) self-injections, in the thigh, of study medication (or have designee perform injection).
9. Willingness and ability to comply with the protocol (prior to screening).
10. With regard to female patients: Women of childbearing potential must have a negative pregnancy test at Screening and agree to use two medically acceptable methods of contraception for the duration of the study with pregnancy testing at every scheduled visit.

EXCLUSION CRITERIA:

Patients who have any of the following during the screening visit are not eligible for enrollment in this study:

1. Known history of hypoparathyroidism resulting from an activating mutation in the CaSR gene or impaired responsiveness to PTH (pseudohypoparathyroidism). If unknown, it shall be assumed to be not-present.
2. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis other than hypoparathyroidism, such as active hyperthyroidism, Paget's disease, insulin-dependent diabetes mellitus (IDDM) or poorly controlled Type II diabetes mellitus (HbA1C > 8%), severe and chronic cardiac, liver or renal disease, Cushing's syndrome, neuromuscular disease such as rheumatoid arthritis, myeloma, pancreatitis, malnutrition, rickets, recent prolonged immobility, active malignancy, primary or secondary hyperparathyroidism, a history of parathyroid carcinoma, hypopituitarism, acromegaly, or multiple endocrine neoplasia types I and II.
3. To be eligible, patients with a history of thyroid cancer must be documented to be disease-free for a period of at least 5 years (or 2 years with evidence of follow up and a doctor's note of clearance).
4. Patients dependent on regular parenteral calcium infusions (e.g. calcium gluconate) to maintain calcium homeostasis.
5. Patients that have undergone gastric resection or have active peptic ulcer disease requiring medical therapy.
6. Use of prohibited medications such as, raloxifene hydrochloride, lithium, methotrexate, or systemic corticosteroids within the last 6 months.
7. Treatment with PTH-like drugs, including PTH(1-84), PTH(1-34) or other N terminal fragments or analogs of PTH or PTH-related protein within the last 6 months.
8. Other drugs known to influence calcium and bone metabolism, such as calcitonin, sodium fluoride, or cinacalcet hydrochloride within the last 6 months.
9. Use of oral bisphosphonates within the previous 6 months or IV bisphosphonate preparations within the previous 12 months prior to screening.
10. Seizure disorder/epilepsy and a history of a documented seizure within the previous 6 months.
11. In regard to participants between 18 and 21 years of age: Presence of open epiphyses as determined by x-ray.
12. Radiotherapy to the skeleton within 5 years.
13. Serum 25-hydroxyvitamin D levels greater than 1.5-fold the laboratory upper limit of normal. (i.e., > 150 ng/mL)
14. Any disease or condition in the opinion of the Investigator that has a high probability of precluding the patient from completing the study or where the patient cannot or will not appropriately comply with study requirements.
15. Participation in any other investigational trial in which receipt of investigational drug or device occurred within 6 months prior to screening for this study.
16. Pregnant or lactating women.
17. History of diagnosed drug or alcohol dependence within the previous 3 years.
18. Clinical history of renal calculi within the past 6 months.
19. Any condition that negatively affects gastrointestinal absorption, including but not limited to short bowel syndrome, bowel resection, tropical sprue, celiac disease, ulcerative colitis, and Crohn's disease.
20. Chronic/severe cardiac disease including but not limited to cardiac insufficiency, arrhythmias, bradycardia (resting heart rate < 60 beats/minute), or hypotension (systolic and diastolic blood pressures < 100 and 60 mmHg, respectively).
21. History of cerebrovascular accident (CVA) in the past 5 years or earlier, if there is residual impairment that would affect participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Bilezikian, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubin MR, Bilezikian JP. Hypoparathyroidism: clinical features, skeletal microstructure and parathyroid hormone replacement. Arq Bras Endocrinol Metabol. 2010 Mar;54(2):220-6. doi: 10.1590/s0004-27302010000200019. PMID 20485912
- [Background] Rubin MR, Sliney J Jr, McMahon DJ, Silverberg SJ, Bilezikian JP. Therapy of hypoparathyroidism with intact parathyroid hormone. Osteoporos Int. 2010 Nov;21(11):1927-34. doi: 10.1007/s00198-009-1149-x. Epub 2010 Jan 22. PMID 20094706
- [Background] Rubin MR, Dempster DW, Kohler T, Stauber M, Zhou H, Shane E, Nickolas T, Stein E, Sliney J Jr, Silverberg SJ, Bilezikian JP, Muller R. Three dimensional cancellous bone structure in hypoparathyroidism. Bone. 2010 Jan;46(1):190-5. doi: 10.1016/j.bone.2009.09.020. Epub 2009 Sep 25. PMID 19782782
- [Background] Rubin MR, Dempster DW, Zhou H, Shane E, Nickolas T, Sliney J Jr, Silverberg SJ, Bilezikian JP. Dynamic and structural properties of the skeleton in hypoparathyroidism. J Bone Miner Res. 2008 Dec;23(12):2018-24. doi: 10.1359/jbmr.080803. PMID 18684087
- [Background] Cusano NE, Rubin MR, Bilezikian JP. PTH(1-84) replacement therapy for the treatment of hypoparathyroidism. Expert Rev Endocrinol Metab. 2015 Jan 1;10(1):5-13. doi: 10.1586/17446651.2015.971755. PMID 25705243
- [Background] Cusano NE, Rubin MR, McMahon DJ, Irani D, Anderson L, Levy E, Bilezikian JP. PTH(1-84) is associated with improved quality of life in hypoparathyroidism through 5 years of therapy. J Clin Endocrinol Metab. 2014 Oct;99(10):3694-9. doi: 10.1210/jc.2014-2267. Epub 2014 Jun 30. PMID 24978675
- [Background] Cusano NE, Rubin MR, Irani D, Sliney J Jr, Bilezikian JP. Use of parathyroid hormone in hypoparathyroidism. J Endocrinol Invest. 2013 Dec;36(11):1121-7. doi: 10.1007/BF03346763. PMID 24445125
- [Background] Cusano NE, Rubin MR, McMahon DJ, Irani D, Tulley A, Sliney J Jr, Bilezikian JP. The effect of PTH(1-84) on quality of life in hypoparathyroidism. J Clin Endocrinol Metab. 2013 Jun;98(6):2356-61. doi: 10.1210/jc.2013-1239. Epub 2013 Apr 17. PMID 23596139
- [Background] Cusano NE, Rubin MR, McMahon DJ, Zhang C, Ives R, Tulley A, Sliney J Jr, Cremers SC, Bilezikian JP. Therapy of hypoparathyroidism with PTH(1-84): a prospective four-year investigation of efficacy and safety. J Clin Endocrinol Metab. 2013 Jan;98(1):137-44. doi: 10.1210/jc.2012-2984. Epub 2012 Nov 15. PMID 23162103
- [Background] Christen P, Ito K, Muller R, Rubin MR, Dempster DW, Bilezikian JP, van Rietbergen B. Patient-specific bone modelling and remodelling simulation of hypoparathyroidism based on human iliac crest biopsies. J Biomech. 2012 Sep 21;45(14):2411-6. doi: 10.1016/j.jbiomech.2012.06.031. Epub 2012 Aug 9. PMID 22883080
- [Background] Cusano NE, Rubin MR, Sliney J Jr, Bilezikian JP. Mini-review: new therapeutic options in hypoparathyroidism. Endocrine. 2012 Jun;41(3):410-4. doi: 10.1007/s12020-012-9618-y. Epub 2012 Feb 7. PMID 22311174
- [Background] Rubin MR, Dempster DW, Sliney J Jr, Zhou H, Nickolas TL, Stein EM, Dworakowski E, Dellabadia M, Ives R, McMahon DJ, Zhang C, Silverberg SJ, Shane E, Cremers S, Bilezikian JP. PTH(1-84) administration reverses abnormal bone-remodeling dynamics and structure in hypoparathyroidism. J Bone Miner Res. 2011 Nov;26(11):2727-36. doi: 10.1002/jbmr.452. PMID 21735476
- [Background] Rubin MR, Manavalan JS, Dempster DW, Shah J, Cremers S, Kousteni S, Zhou H, McMahon DJ, Kode A, Sliney J, Shane E, Silverberg SJ, Bilezikian JP. Parathyroid hormone stimulates circulating osteogenic cells in hypoparathyroidism. J Clin Endocrinol Metab. 2011 Jan;96(1):176-86. doi: 10.1210/jc.2009-2682. Epub 2010 Sep 29. PMID 20881259
- [Derived] Ayodele O, Rejnmark L, Mu F, Lax A, Berman R, Swallow E, Gosmanova EO. Five-Year Estimated Glomerular Filtration Rate in Adults with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Nov;39(11):5013-5024. doi: 10.1007/s12325-022-02292-1. Epub 2022 Aug 26. PMID 36018496
- See also: The Hypoparathyroidism Association — http://hypoPARA.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label PTH(1-84)
Started | 62
Completed (At 4 years) | 27
Completed (At study conclusion) | 13
Not Completed | 49

BASELINE CHARACTERISTICS:
Arm/Group | Open-label PTH(1-84)
Number analyzed (Participants) | 62
Age, Customized [Count of Participants; unit: Participants]
  18-21 years | 0
  22-29 years | 5
  30-39 years | 7
  40-49 years | 22
  50-59 years | 13
  60-69 years | 13
  70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Dose of Calcium Supplementation
Description: Serum and urinary calcium levels maintained by change in requirements for calcium supplementation.
Time Frame: Baseline, up to 4 years
Population: Analyzed data from this cohort included 27 evaluable subjects treated with open-label PTH(1-84) for 4 years.
Measure: Mean (Standard Deviation); unit: percent change in dose
Arm/Group | Open-label PTH(1-84)
Number analyzed (Participants) | 27
percent change in dose | 37 (43)

2. Secondary Outcome: Percent Change in BMD by DXA
Description: Bone Mineral Density (BMD) as measured by Dual Energy X-Ray Absorptiometry (DXA)
Time Frame: Baseline, up to 4 years
Population: Analyzed data from this cohort included 27 evaluable subjects treated with open-label PTH(1-84) for 4 years.
Measure: Mean (Standard Deviation); unit: percent change in BMD
Arm/Group | Open-label PTH(1-84)
Number analyzed (Participants) | 27
percent change in BMD | 5.5 (9)

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Arm/Group | Open-label PTH(1-84)
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 25/62
Other Adverse Events (participants affected / at risk) | 27/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label PTH(1-84) (N=62)
Hypercalcemia (Endocrine disorders) | 1 (1)
Hypocalcemia (Endocrine disorders) | 13 (13)
Pneumonia (Infections and infestations) | 2 (2)
Surgery elective (Surgical and medical procedures) | 3 (3)
Swelling of face, tongue (Endocrine disorders) | 3 (3)
Gastroenteretis (Gastrointestinal disorders) | 1 (1)
Infection in uterus (Reproductive system and breast disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label PTH(1-84) (N=62)
Muscular/skeletal event (Musculoskeletal and connective tissue disorders) | 16
Circulatory event (Vascular disorders) | 4
Digestive event (Gastrointestinal disorders) | 5
Endocrine/Nutritional event (Endocrine disorders) | 9
Infection (General disorders) | 8
Nervous system event (Nervous system disorders) | 5
Urinary event (Renal and urinary disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT01199614/Prot_SAP_000.pdf